CLINICAL TRIAL: NCT05250180
Title: Using Dogs to Promote Therapeutic Engagement During Inpatient Rehabilitation Following Pediatric Acquired Brain Injury: Understanding Mechanisms and Moderators of Treatment Response.
Brief Title: Animal Assisted Therapy After Pediatric Brain Injury: Mediators and Moderators of Treatment Response.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Miami University (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Cin AAT for ABI; 1R01HD106416 (NIH)
Record Dates: First submitted 2022-01-21; First posted 2022-02-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Brain Injuries
Keywords: Pediatric brain injury; Animal assisted therapy; inpatient rehabilitation
MeSH Terms: conditions — Brain Injuries | interventions — Animal Assisted Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): animal assisted therapy
  Interventions: Other: Animal Assisted Therapy
- Control (Active Comparator): Treatment as usual
  Interventions: Other: Control

INTERVENTIONS:
Other: Animal Assisted Therapy — Patients enrolled in the study will be randomly scheduled to have a dog be a part of their PT and OT sessions on two days (one in the first week and one in the second week) during their stay. On these days, the therapist will lead the therapy session and integrate the dog at whatever level is appropriate based on the patient's level of functioning and therapy goals.
  Other Names: AAT
  Arms: Intervention
Other: Control — treatment as usual as dictated by their treatment team
  Other Names: Treatment as usual
  Arms: Control

SUMMARY:
Children requiring inpatient rehabilitation treatment following acquired brain injury (ABI) are at risk for poor engagement in rehabilitative therapies. A within subject crossover design will be used to determine whether involving dogs in physical and occupational therapies while receiving inpatient rehabilitation improves patient engagement, how involving dogs improves engagement, and identify who is most likely to benefit. This project addresses the critical need to establish an evidence base for animal-assisted therapies in pediatric rehabilitation, incorporates innovative methods, and has the potential to lead to improved clinical care for children and adolescents receiving intensive rehabilitation following ABI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Participants must be admitted to the inpatient rehabilitation unit for treatment of an acquired brain injury (TBI, brain tumor, infection, etc).
* Consent: The family must provide informed consent by parents or legal guardians.
* Assent: The child/adolescent must provide a signature indicating assent to participate in the study.
* Age at the time of screening: 4-21 years old
* Sex: includes both males and females
* Responsiveness: Rancho score greater than 2 at the time of enrollment (as noted in the medical chart).

Exclusion Criteria:

* Allergies: Patient has a significant allergy to dogs
* Fear: Patient has a significant fear of dogs
* Disease: Participant is on contact precautions or has a communicable disease that may pose a risk to the dog or dog handler or has a compromised immune system where interacting with the dog and/or handler would be of significant risk to the patient.
* Medical History: History of developmental delay prior to ABI.
* Behavioral History: Participant or family has a history of animal abuse or cruelty.
* Responsiveness: Rancho score of 2 or less

Ages: 4 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Participation/engagement | throughout study completion - an average of 2 weeks
  Patient engagement/participation will be assessed via the Pittsburgh Rehabilitation Participation Scale (PRPS) is a 6-item Likert-type, clinician-rated measure that quantifies observed patient participation/engagement in their therapy sessions. Therapists will report their observations regarding patient's completion of exercises, effort applied to exercises, and level of support needed to complete activities.
Objective Engagement rating. | throughout study completion - an average of 2 weeks
  An objective measure of session engagement assessed via behavioral coding of video recorded therapy sessions. Coders will provide an objective measure of engagement by rating the patient in-session engagement based on the PRPS. Behaviors reflective of ratings on the PRPS will be clearly operationalized with anchors for each rating clearly defined.

SECONDARY OUTCOMES:
Patient-reported mood | throughout study completion - an average of 2 weeks
  Symptom Inventory Short form is a 4-item scale that asks participants to rate their level of happiness, fatigue, distraction, and irritability on a scale from 1-10.
Objective mood assessment | throughout study completion - an average of 2 weeks
  Objective mood assessment will be completed via behavioral coding of session videos using Noldus Observer software. Coders will code six overarching constructs - Positive affect, negative affect, anxious-fearful affect, neutral affect, touch-physical contact, and persistence on task - with clearly defined and operationalized behaviors that contribute to each construct.
Automated mood assessment | throughout study completion - an average of 2 weeks
  Automated mood assessment will be completed using Noldus FaceReader software. FaceReader is a robust automated system for the recognition of a number of specific properties in facial images, including a neutral state as well as the six basic or universal expressions - happy, sad, angry, surprised, scared, and disgusted.
Physiological distress | throughout study completion - an average of 2 weeks
  Physiological variables - electrodermal activity, heart rate, and heart rate variability - will be collected continuously throughout each therapy session via Empatica E4 wristband. The average electrodermal activity, mean heart rate, heart rate variability (RMSSD: Square root of the mean squared differences of successive intervals) will be used as indicators of physiological distress during sessions.
Salivary Oxytocin | throughout study completion - an average of 2 weeks
  Level of oxytocin present in patient's saliva

OTHER OUTCOMES:
Anthropomorphism | throughout study completion - an average of 2 weeks
  Anthropomorphism is the tendency to attribute human like characteristics, particularly internal states and capabilities, to non-human entities. Patient level of anthropomorphism will be assessed via the 12-item Individual Differences in Anthropomorphism Questionnaire - Child Form.
Patient-animal rapport | throughout study completion - an average of 2 weeks
  patient-animal rapport will be assessed via the patient-animal closeness measure. Patients are presented with 7 images and asked to select a number between 1 and 7 that best describes the amount of overlap between the patient and the dog.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States